CLINICAL TRIAL: NCT04129671
Title: Rare Variation and Remote Gene Regulation of Osteoporosis Related Phenotypes in Han Chinesse
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Westlake University (Other)
Responsible Party: Principal Investigator, Shigui Yan, Honorary director of the department of orthopaedics surgery, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: 2018-090
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Senile Osteoporosis With Current Pathological Fracture Lower Leg (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from whole blood samples of the patients with osteoporosis fractures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: No intervention was applied — No intervention was administered

SUMMARY:
Bone density is recognized as the most important factor to measure osteoporosis, and the prevalence of osteoporosis increases with age. Risk factors for osteoporosis include age, weight, exercise, diet, smoking and alcohol consumption. What's more, osteoporosis has a strong familial aggregation, and the genetic value of bone density is between 0.6 and 0.85. Therefore, it is necessary to conduct large-scale collection of population samples of osteoporosis fractures and relevant genetic studies.

DETAILED DESCRIPTION:
From past linkage analysis and candidate gene association studies to genome-wide association studies and second-generation sequencing technologies, researchers have found hundreds of genes and SNPs associated with bone mineral density and osteoporosis fractures. However, current studies on osteoporosis and related phenotypes are mainly concentrated in the European and American populations, rare in Asia and other regions, and even less in the Chinese han population. It is one of the problems to be solved in this project whether the genes and SNP loci associated with these strengths can also be applied to han Chinese population due to the existence of racial differences. This project aims to collect the patients with primary osteoporosis and osteoporosis fracture in the Chinese han population through the orthopaedics department, and verify the identified osteoporosis susceptibility genes in the Chinese han population.

ELIGIBILITY:
Inclusion Criteria:

1. From July 2018 to July 2021, patients admitted to the outpatient or inpatient clinic were diagnosed as primary osteoporosis fracture;
2. Aged between 50 and 100;
3. This fracture was not treated with any anti-osteoporosis drugs before
4. Subjects will participate in the study voluntarily and have signed the informed consent
5. Patients with clear mind and independent behavioral ability

Exclusion Criteria:

1. Patients with malignant tumors are associated with bone metastases, such as lung cancer, prostate cancer, thyroid cancer, etc
2. Hyperparathyroidism, Cushing syndrome, hypogonadism, hyperthyroidism, pituitary prolactinoma, diabetes
3. Systemic lupus erythematosus, rheumatoid arthritis, sjogren's syndrome, dermatomyositis, mixed connective tissue disease, etc.;
4. Renal osteodystrophy caused by various chronic kidney diseases;
5. Gastrointestinal diseases and nutritional diseases: malabsorption syndrome, subtotal gastrectomy, chronic pancreatic diseases, chronic liver diseases, protein-calorie malnutrition, long-term intravenous nutrition support treatment, etc.;
6. Leukemia, lymphoma, multiple myeloma, hyperthermia and myelodysplastic syndrome;
7. Hemiplegia, paraplegia, motor dysfunction, muscular dystrophy, catalepsy and myotonic syndrome caused by various reasons;
8. Glucocorticoids, immunosuppressants, heparin, anticonvulsants, anticancer drugs, aluminum-containing antacids, thyroid hormones, gnrh-a or dialysate, etc.
9. Unwilling to accept dietary management or unable to sign the informed consent

Ages: 50 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. From July 2018 to July 2021, patients admitted to the outpatient or inpatient clinic were diagnosed as primary osteoporosis fracture;
  2. Aged between 50 and 100;
  3. This fracture was not treated with any anti-osteoporosis drugs before
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Exon sequencing results from the target region | June 2018-December 2021
  Exon sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejing Province, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] He W, Liu M, Huang X, Qing Z, Gao W. The influence of vitamin D receptor genetic variants on bone mineral density and osteoporosis in Chinese postmenopausal women. Dis Markers. 2015;2015:760313. doi: 10.1155/2015/760313. Epub 2015 Feb 17. PMID 25784778
- [Result] Mendoza N, Quereda F, Presa J, Salamanca A, Sanchez-Borrego R, Vazquez F, Martinez Astorquiza T. Estrogen-related genes and postmenopausal osteoporosis risk. Climacteric. 2012 Dec;15(6):587-93. doi: 10.3109/13697137.2012.656160. Epub 2012 Feb 15. PMID 22335445